CLINICAL TRIAL: NCT00117741
Title: Evaluation of Dialectical Behavior Therapy (DBT)
Brief Title: Evaluation of DBT Compared to Drug Counseling for Opiate Addicts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Marsha Linehan, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DA014997 (NIH); R01DA014997 (NIH)
Record Dates: First submitted 2005-06-30; First posted 2005-07-08 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Opiate Addiction; Borderline Personality Disorder
Keywords: Opiate Dependence; DBT; Dialectical Behavior Therapy; Drug Counseling; Therapy, Cognitive Behavior
MeSH Terms: conditions — Opioid-Related Disorders; Borderline Personality Disorder | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dialectical Behavior Therapy (Experimental): Participants receive standard dialectical behavior therapy and suboxone
  Interventions: Behavioral: Dialectical Behavior Therapy
- Drug Counseling (Active Comparator): Participants receive standard individual and group counseling and suboxone.
  Interventions: Behavioral: Drug Counseling

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy — Weekly individual DBT, DBT group skills training, as needed phone calls for coaching, team meeting for psychotherapists, suboxone
  Other Names: DBT
  Arms: Dialectical Behavior Therapy
Behavioral: Drug Counseling — Weekly individual counseling and weekly group therapy following guidelines of drug counseling treatment manual,
  Other Names: Individual and Group Drug Counseling
  Arms: Drug Counseling

SUMMARY:
The purpose of this study is to compare a one year treatment program of Dialectical Behavior Therapy (DBT) + suboxone for opiate addicted individuals meeting criteria for borderline personality disorder (BPD) to a one year program of standard drug counseling (I/GDC) + suboxone.

DETAILED DESCRIPTION:
The purpose of this study is to compare a one year treatment program of Dialectical Behavior Therapy (DBT) + suboxone for opiate addicted individuals meeting criteria for borderline personality disorder (BPD) to a one year program of standard drug counseling (I/GDC) + suboxone. Drug counseling consists of manualized individual sessions + group therapy. This trial is being completed at two sites, at the University of Washington and at Duke University. One hundred and seventy-two individuals (86 per condition) with opiate dependence and meeting criteria for BPD will be enrolled in a one-year treatment and a one-year follow-up assessment. Each site (University of Washington, Duke) will enroll 86 clients with both treatment conditions being conducted at each site. Assessments measuring drug use, suicidal behaviors, retention and other treatment-related behaviors, general psychopathology and functioning, and increases in behavioral skills will be given at four month intervals for the entire two years.

ELIGIBILITY:
Inclusion Criteria:

* 1. Meets SCID-I criteria for opiate dependence. 2. Meets IPDE and SCID criteria for BPD (DSM-IV) 3. Over 18 years old 4. Resides within commuting distance of treatment 5. Consents to outpatient treatment for drug addiction

Exclusion Criteria:

* 1. Bipolar, Schizophrenia, Schizophreniform, or Schizoaffective Disorders, Psychosis NOS 2. IQ less than 70; life threatening anorexia; current and chronic absence of shelter; impending jail/prison for more than three weeks (problems which by their presence or severity preclude ability to attend or understand treatment and/or requires priority treatment over SUD treatment) 3. Court order to treatment, court order to treatment or to jail, or agency order to treatment or loss of child custody (due to consequent inability to freely drop-out of treatment) 4. Is pregnant, plans to become pregnant during treatment phase, or becomes pregnant before random assignment to study condition 5. Is unable to tolerate suboxone induction phase 6. Is currently stable on methadone 7. Current benzodiazepine use from which the participant is unwilling to taper 8. Refuses: to discontinue current mental health or drug abuse treatment or random assignment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2004-06; Primary Completion 2008-10 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Urinalysis | one year treatment, one year follow-up

SECONDARY OUTCOMES:
Suicidal Behavior | one year treatment, one year follow-up
Depression, anxiety, Axis I diagnostic remission | one year treatment, one year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Marsha Linehan, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Behavioral Research and Therapy Clinics, Seattle, Washington, United States

REFERENCES:
- [Background] Linehan MM, Armstrong HE, Suarez A, Allmon D, Heard HL. Cognitive-behavioral treatment of chronically parasuicidal borderline patients. Arch Gen Psychiatry. 1991 Dec;48(12):1060-4. doi: 10.1001/archpsyc.1991.01810360024003. PMID 1845222
- [Background] Linehan MM, Tutek DA, Heard HL, Armstrong HE. Interpersonal outcome of cognitive behavioral treatment for chronically suicidal borderline patients. Am J Psychiatry. 1994 Dec;151(12):1771-6. doi: 10.1176/ajp.151.12.1771. PMID 7977884
- [Background] Linehan MM, Dimeff LA, Reynolds SK, Comtois KA, Welch SS, Heagerty P, Kivlahan DR. Dialectical behavior therapy versus comprehensive validation therapy plus 12-step for the treatment of opioid dependent women meeting criteria for borderline personality disorder. Drug Alcohol Depend. 2002 Jun 1;67(1):13-26. doi: 10.1016/s0376-8716(02)00011-x. PMID 12062776
- [Background] Linehan MM, Schmidt H 3rd, Dimeff LA, Craft JC, Kanter J, Comtois KA. Dialectical behavior therapy for patients with borderline personality disorder and drug-dependence. Am J Addict. 1999 Fall;8(4):279-92. doi: 10.1080/105504999305686. PMID 10598211
- [Background] Verheul R, Van Den Bosch LM, Koeter MW, De Ridder MA, Stijnen T, Van Den Brink W. Dialectical behaviour therapy for women with borderline personality disorder: 12-month, randomised clinical trial in The Netherlands. Br J Psychiatry. 2003 Feb;182:135-40. doi: 10.1192/bjp.182.2.135. PMID 12562741
- See also: Click here for more information about the Behavioral Research and Therapy Clinics at the University of Washington — http://depts.washington.edu/brtc/